CLINICAL TRIAL: NCT03869957
Title: Effect of Parenteral Nutrition With n-3 PUFAs on Patients With Intestinal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Aurora Elizabeth Serralde Zúñiga, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2846
Record Dates: First submitted 2019-02-25; First posted 2019-03-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Intestinal Failure
Keywords: omega 3 polyunsaturated fatty acids; intestinal failure; oxidative stress
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: A team researcher will use Stata 12, to perform randomization with a 1:1 allocation using random block sizes of 4. Once the treatment group is determined, the PN will be prescribed accordingly and the preparation will be carried out in the pharmacy and it will have the same appearance in both arms. Patients and researchers who will evaluate the outcomes and perform the statistical analysis will be blinded to the assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): We will use ~0.8-0.9 g/kg/day of Clinoleic® (80% olive oil/20 soybean oil) + 0.2-0.1 g/kg/day [Omegaven® ](100% fish oil), to cover the proposed amount of n-3 PUFAs for 7 days. The infusion rate should not exceed 0.5 ml Omegaven® / kg body weight / hour = 0.05 g fish oil / kg body weight / hour. The intervention group will return to PN without n-3 PUFA after 7 days.
  Interventions: Dietary Supplement: Intervention group
- Control group (No Intervention): Will be administering ~1.0 g/kg/d the lipid emulsion Clinoleic® (80% olive oil/20 soybean oil) without n-3 PUFAs.

INTERVENTIONS:
Dietary Supplement: Intervention group — 0.1-0.2 g n-3 PUFA/kg body weight/day for 7 days
  Other Names: n-3 PUFAs
  Arms: Intervention group

SUMMARY:
Randomized, double-blind, controlled clinical trial to evaluate the effect of parenteral nutrition (PN) supplemented with lipid emulsions containing 0.1-0.2 g omega 3 polyunsaturated fatty acids (n-3 PUFA)/kg body weight/day for 7 days on malondialdehyde (MDA) levels, a marker of lipoperoxidation of reactive species, compared with a control group (without n-3 PUFA) in patients with intestinal failure (IF).

DETAILED DESCRIPTION:
IF is the loss of intestinal function that affects the decrease in the absorption of macronutrients, water, and electrolytes, so it requires intravenous supplementation such as PN and/or intravenous fluids to maintain health and/or growth. IF type II is associated with complex infectious and metabolic complications and patients require PN for weeks or months. Long-term PN use, however, includes the risk of complications, among which a serious one is the intestinal failure-associated liver disease (1). It has been proposed that metabolic endotoxemia (2-3), inflammation (4) and oxidative stress (5) are involved in the development of this intestinal failure-associated liver disease.

Although some studies have reported beneficial effects of n-3 PUFA to prevent and reverse the liver disease associated with IF (6-7), due to its antioxidant (8-10) and anti-inflammatory activity (11-12) and in the modulation of the intestinal microbiota (13), the literature on the use of n-3 PUFA in non-critical patients with IF and PN is limited and the results have not been conclusive.

Therefore, a randomized, double-blind, controlled clinical trial to evaluate the effect of PN supplemented with lipid emulsions containing n-3 PUFA/kg body weight/day for 7 days on oxidative stress (concentrations of MDA), compared with a control group (without n-3 PUFA) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the non-critical areas of the Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ) with a nutritional risk between January 2019 and July 2020 will be considered eligible.
* Patients with recent diagnosis of IF type II (an evolution >28 days) originate from various gastrointestinal or systemic diseases (short bowel, intestinal fistula, intestinal dysmotility, mechanical obstruction, and extensive small bowel mucosal disease).

Exclusion Criteria:

* Patients with contraindications for PN
* Patients with known allergies to the components of the PN formula
* Severe liver or renal insufficiency
* Uncontrolled diabetes mellitus
* Certain acute and life-threatening conditions
* Immunological diseases (such as autoimmune diseases, human immunodeficiency virus infection, cancer, etc.)
* Those that take immunosuppressant medications
* Severe hemorrhagic disorders
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change of malondialdehyde (MDA) in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Measurement of malondialdehyde (MDA) that is a marker for oxidative stress, determined in serum in ng/dl.

SECONDARY OUTCOMES:
Change of glutathione (GSH) in plasma from baseline to day 7 | Change from baseline (day 0) at day 7
  Measurement of glutathione (GSH) that is a marker for oxidative stress, determined in plasma in micromol/l.
Change of oxidized glutathione (GSSG) in plasma from baseline to day 7 | Change from baseline (day 0) at day 7
  Measurement of oxidized glutathione (GSSG) that is a marker for oxidative stress, determined in plasma in micromol/l.
Change of GSH/GSSG ratio from baseline to day 7 | Change from baseline (day 0) at day 7
  GSH and GSSG will be combined to report GSH/GSSG ratio in micromol/l
Change of carbonylated protein in serum from baseline to day 7. | Change from day 0 at day 7.
  Measurement of carbonylated protein that is a marker for oxidative stress, determined in serum in nmol/mg
Change of lipopolysaccharide (LPS) in serum from baseline to day 7. | Change from baseline (day 0) at day 7
  Measurement of lipopolysaccharide (LPS) that is a marker for metabolic endotoxemia, determined in serum in ng/dl.
Change of C-reactive protein (CRP) in serum from baseline to day 7. | Change from baseline (day 0) at day 7
  Measurement of C-reactive protein (CRP) that is a marker for inflammation, determined in serum in pg/ml.
Change of glucose in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of glucose in serum according medical records, in mg/dl
Change of nitrogen ureic in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of nitrogen ureic in serum according medical records, in mg/dl
Change of urea in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of urea in serum according medical records, in mg/dl
Change of creatinin in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of creatinin in serum according medical records, in mg/dl
Change of sodium in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of sodium in serum according medical records, in mmol/l
Change of potassium in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of potassium in serum according medical records, in mmol/l
Change of phosphorus in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of phosphorus in serum according medical records, in mg/dl
Change of magnesium in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of magnesium in serum according medical records, in mg/dl
Change of total bilirubin in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of total bilirubin in serum according medical records, in mg/dl
Change of direct bilirubin in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of direct bilirubin in serum according medical records, in mg/dl
Change of indirect bilirubin in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of indirect bilirubin in serum according medical records, in mg/dl
Change of alanine aminotransferase in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of alanine aminotransferase in serum according medical records, in U/l
Change of aspartate aminotransferase in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of aspartate aminotransferase in serum according medical records, in U/l
Change of alkaline phosphatase in serum from baseline to day 7 | Change from baseline (day 0) at day 7
  Concentration of alkaline phosphatase in serum according medical records, in U/l
Frequency of patients with nutritional risk at baseline | At baseline (day 0)
  Determine the frequency of patients with nutritional risk according the Nutritional Risk Assesment-2002 (NRS-2002) tool, in percentage.
Determine the type of intestinal failure at baseline. | At baseline (day 0)
  Identify the classification of patients with intestinal failure according the ESPEN guidelines on chronic intestinal failure in adults, in percentage.
Frequency of primary diagnosis at baseline. | At baseline (day 0)
  Determine the frequency of primary diagnosis according medical records, in percentage.
Assessment of resting energy expenditure at baseline | Baseline (day 0)
  Measurement of resting energy expenditure at baseline with a calorimeter, in kcal/day
Assessment of nutritional prescription at baseline and at day 7 | At baseline (day 0) and at day 7
  Determine the nutritional prescription at baseline, in kcal/day
Frequency of the type and characteristics of nutritional support administered | At baseline (day 0) and at day 7
  Determine type and characteristics of nutritional support administered, according medical records, in percentage
Assessment of height at baseline | Baseline (day 0)
  Measurement of weight in centimeters
Assessment of weight at baseline and at the end of the follow-up | At baseline (day 0) and at the end of the follow-up (~ at day 30)
  Measurement of weight in kilograms
Assessment of body mass index at baseline and at the end of the follow-up | At baseline (day 0) and at the end of the follow-up (~ at day 30)
  Weight and height will be combined to report BMI in kg/m^2
Assessment of percentage of lean mass at baseline and at the end of the follow-up | At baseline (day 0) and at the end of the follow-up (~ at day 30)
  Measurement of percentage of lean mass at baseline with a electric bioimpedance (InBody S10 ®).
Assessment of percentage of fat mass at baseline and at the end of the follow-up | At baseline (day 0) and at the end of the follow-up (~ at day 30)
  Measurement of percentage of fat mass at baseline with a electric bioimpedance (InBody S10 ®).
Assessment of muscle function at baseline and at the end of the follow-up | At baseline (day 0) and at the end of the follow-up (~ at day 30)
  Measurement of muscle function with a handgrip at baseline, in kilograms
Length of stay at hospitalization area | From the date of admission to the date of discharge from the hospitalization area (~ at day 30)
  Determine the length of stay from the date of admission to the date of discharge from the hospitalization area, in days
Rate of mortality | At the end of the follow-up (~ at day 30)
  Evaluation of frequency of mortality, in percentage
Frequency of intestinal failure-associated liver disease (IFALD) | From baseline (day 0) to the end of the follow-up (~ at day 30)
  Determined with the elevation in alkaline phosphatase concentrations within the first 7-14 days with parenteral nutrition, by elevation in transaminase concentrations more than 1.5 times above the upper limit of reference, or by elevation in the total bilirubin or direct bilirubin concentrations >3, 4, 6 and 12 mg / dl
Change in lipidomics in serum from day 0 to day 7 | Change from baseline (day 0) to day 7
  Change in lipidomic profile of the diferent lipid species

CONTACTS AND LOCATIONS:
Overall Officials: Aurora E Serralde-Zúñiga, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

REFERENCES:
- [Result] Pironi L, Arends J, Baxter J, Bozzetti F, Pelaez RB, Cuerda C, Forbes A, Gabe S, Gillanders L, Holst M, Jeppesen PB, Joly F, Kelly D, Klek S, Irtun O, Olde Damink SW, Panisic M, Rasmussen HH, Staun M, Szczepanek K, Van Gossum A, Wanten G, Schneider SM, Shaffer J; Home Artificial Nutrition & Chronic Intestinal Failure; Acute Intestinal Failure Special Interest Groups of ESPEN. ESPEN endorsed recommendations. Definition and classification of intestinal failure in adults. Clin Nutr. 2015 Apr;34(2):171-80. doi: 10.1016/j.clnu.2014.08.017. Epub 2014 Sep 21. PMID 25311444
- [Result] Korpela K, Mutanen A, Salonen A, Savilahti E, de Vos WM, Pakarinen MP. Intestinal Microbiota Signatures Associated With Histological Liver Steatosis in Pediatric-Onset Intestinal Failure. JPEN J Parenter Enteral Nutr. 2017 Feb;41(2):238-248. doi: 10.1177/0148607115584388. Epub 2016 Sep 30. PMID 25934046
- [Result] Omata J, Pierre JF, Heneghan AF, Tsao FH, Sano Y, Jonker MA, Kudsk KA. Parenteral nutrition suppresses the bactericidal response of the small intestine. Surgery. 2013 Jan;153(1):17-24. doi: 10.1016/j.surg.2012.04.001. Epub 2012 Jun 13. PMID 22698933
- [Result] Cadenas S, Cadenas AM. Fighting the stranger-antioxidant protection against endotoxin toxicity. Toxicology. 2002 Oct 30;180(1):45-63. doi: 10.1016/s0300-483x(02)00381-5. PMID 12324199
- [Result] Lacaille F, Gupte G, Colomb V, D'Antiga L, Hartman C, Hojsak I, Kolacek S, Puntis J, Shamir R; ESPGHAN Working Group of Intestinal Failure and Intestinal Transplantation. Intestinal failure-associated liver disease: a position paper of the ESPGHAN Working Group of Intestinal Failure and Intestinal Transplantation. J Pediatr Gastroenterol Nutr. 2015 Feb;60(2):272-83. doi: 10.1097/MPG.0000000000000586. PMID 25272324
- [Result] Nandivada P, Fell GL, Gura KM, Puder M. Lipid emulsions in the treatment and prevention of parenteral nutrition-associated liver disease in infants and children. Am J Clin Nutr. 2016 Feb;103(2):629S-34S. doi: 10.3945/ajcn.114.103986. Epub 2016 Jan 20. PMID 26791189
- [Result] Burns DL, Gill BM. Reversal of parenteral nutrition-associated liver disease with a fish oil-based lipid emulsion (Omegaven) in an adult dependent on home parenteral nutrition. JPEN J Parenter Enteral Nutr. 2013 Mar;37(2):274-80. doi: 10.1177/0148607112450301. Epub 2012 Jun 8. PMID 22683685
- [Result] Ventro G, Chen M, Yang Y, Harmon CM. Molecular impact of omega 3 fatty acids on lipopolysaccharide-mediated liver damage. J Pediatr Surg. 2016 Jun;51(6):1039-43. doi: 10.1016/j.jpedsurg.2016.02.078. Epub 2016 Mar 2. PMID 27072665
- [Result] Wu G, Zhou W, Zhao J, Pan X, Sun Y, Xu H, Shi P, Geng C, Gao L, Tian X. Matrine alleviates lipopolysaccharide-induced intestinal inflammation and oxidative stress via CCR7 signal. Oncotarget. 2017 Feb 14;8(7):11621-11628. doi: 10.18632/oncotarget.14598. PMID 28086227
- [Result] Giordano E, Visioli F. Long-chain omega 3 fatty acids: molecular bases of potential antioxidant actions. Prostaglandins Leukot Essent Fatty Acids. 2014 Jan;90(1):1-4. doi: 10.1016/j.plefa.2013.11.002. Epub 2013 Dec 3. PMID 24345866
- [Result] Calder PC. Omega-3 fatty acids and inflammatory processes: from molecules to man. Biochem Soc Trans. 2017 Oct 15;45(5):1105-1115. doi: 10.1042/BST20160474. Epub 2017 Sep 12. PMID 28900017
- [Result] Osowska S, Kunecki M, Sobocki J, Tokarczyk J, Majewska K, Omidi M, Radkowski M, Fisk HL, Calder PC. Effect of changing the lipid component of home parenteral nutrition in adults. Clin Nutr. 2019 Jun;38(3):1355-1361. doi: 10.1016/j.clnu.2018.05.028. Epub 2018 Jun 6. PMID 29907355
- [Result] Laparra JM, Sanz Y. Interactions of gut microbiota with functional food components and nutraceuticals. Pharmacol Res. 2010 Mar;61(3):219-25. doi: 10.1016/j.phrs.2009.11.001. Epub 2009 Nov 13. PMID 19914380